CLINICAL TRIAL: NCT00286962
Title: A Randomized Cross-Over Single Centre Study Comparing the Effects of Intraperitoneal Insulin Administration to Subcutaneous Insulin Administration in Type 1 Diabetes Mellitus Patients
Brief Title: Study to Compare Intraperitoneal Insulin to Subcutaneous Insulin Administration in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Foundation, The Netherlands (Other)
Collaborators: Medtronic (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IC-06-01-SL; 04.0211p
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes mellitus, type 1; insulin infusion systems; continuous intraperitoneal insulin infusion; cross-over studies
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- CIPII (Experimental): Intraperitoneal insulin infusion by means of an implanted insulin pump
  Interventions: Device: MIP 2007C implantable insulin pump
- CSII/ MDI (Active Comparator): Optimized subcutaneous insulin infusion by means of continuous subcutaneous insulin infusion (CSII) or by multiple daily injections (MDI)
  Interventions: Device: continuous subcutaneous insulin infusion (CSII) or MDI

INTERVENTIONS:
Device: MIP 2007C implantable insulin pump — Intraperitoneal insulin infusion delivered by an implantable pump: MIP 2007c
  Arms: CIPII
Device: continuous subcutaneous insulin infusion (CSII) or MDI
  Arms: CSII/ MDI

SUMMARY:
The purpose of this study is to compare intraperitoneal (IP) therapy to subcutaneous administration of insulin regarding safety, glycemic control and number of episodes of hypoglycemia in patients with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Various study data available suggest that intraperitoneal (IP) delivery of insulin in type 1 and type 2 diabetic subjects provides an appropriate therapy that allows subjects to achieve acceptable glycemic control without increasing the inherent risk of severe hypoglycemia observed when intensive insulin treatment is pursued. Up till now little research has been done to investigate the efficacy of intraperitoneal (IP) therapy compared to subcutaneous administration. In this study we aim for safety and non-inferiority or superiority for IP therapy concerning glycemic control with less episodes of hypoglycemia compared to intensive subcutaneous (SC) therapy in intermediate or poorly controlled Type 1 patients and/or patients with frequent severe hypoglycemic events.

Subjects will be randomized to insulin treatment using the Medtronic Minimed Implantable Pump or to subcutaneous insulin therapy during the first study arm. After the first arm of the study, subjects will be crossed over to the second arm and will receive the treatment whichever they had not received in the first treatment phase. Subjects with the MIP already implanted will retain the pump but will receive diluent intraperitoneally for the second study arm.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus
* Intermediate or poor glycemic control, defined as HbA1c ≥ 7,5% AND/OR ≥ 5 incidents of hypoglycemia a week.

Exclusion Criteria:

* renal function impairment: creatinin ≥ 150 micromol/L or a creatinin clearance < 50 ml/min
* Cardiac problems: decompensated heart failure (NYHA III and IV); diagnosis of unstable angina pectoris; myocardial infarction within the last 12 months
* Known or suspected allergy against insulin or any component of the composition
* Mental retardation or psychiatric treatment for schizophrenia, organic mental disorder or bipolar disorder currently or in the past.
* Severe untreated proliferative retinopathy.
* Insufficient knowledge of the Dutch language to understand the requirements of the study.
* Current use of systemic corticosteroids or suffering from a condition which caused systemic corticosteroid use more than once in the last year.
* Substance abuse, other than nicotine
* A history of cancer, excluding well differentiated thyroid carcinoma, breast carcinoma without lymph node metastases and skin carcinoma
* Participation in other trials, involving investigational products within 30 days prior to trial entry.
* Plans to engage in activities which require them to go below 25 feet below sea level.
* Any condition that the Investigator and/or Coordinating Investigator feels would interfere with trial participation or evaluation of results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
incidence of hypoglycemia; data taken from patient diaries during either study arm.

SECONDARY OUTCOMES:
glycemic control; glycosylated hemoglobin (HbA1c) measurement at baseline, end of entry phase, start of both study arms, halfway through study arms, end of study arms.
average daily insulin usage; as taken from patient diaries for both study arms
frequency of adverse events; as taken from patient diaries for both study arms
frequency of clinically significant abnormal laboratory values and device complications; as taken from patient diaries for both study arms
Quality of life; score on a quality of life scale at baseline and end of either study arm
Treatment satisfaction; score on treatment satisfaction scale at baseline and end of either study arm
daily glucose excursions; measured with continuous glucose monitoring system (CGMS) at baseline, halfway through and at the end of both study arms

CONTACTS AND LOCATIONS:
Overall Officials: Henk J Bilo, MD, PhD, Principal Investigator — Isala Clinics, medical research foundation
Locations (1):
- Isala Klinieken, Zwolle, Netherlands

REFERENCES:
- [Derived] Logtenberg SJ, Kleefstra N, Houweling ST, Groenier KH, Gans RO, Bilo HJ. Health-related quality of life, treatment satisfaction, and costs associated with intraperitoneal versus subcutaneous insulin administration in type 1 diabetes: a randomized controlled trial. Diabetes Care. 2010 Jun;33(6):1169-72. doi: 10.2337/dc09-1758. Epub 2010 Feb 25. PMID 20185731